CLINICAL TRIAL: NCT02514928
Title: Resection of the Nerve Plexus on the Right Half of Celiac and SMA Associated With Extended Pancreatoduodenectomy in the Surgical Treatment for Adenocarcinoma of the Head of Pancreas
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PCI003
Record Dates: First submitted 2015-08-02; First posted 2015-08-04 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pancreatoduodenectomy & nerve resection (Experimental): Resection of the nerve plexus on the right half of celiac and SMA associated with extended pancreatoduodenectomy. Regional lymph nodes includes group 5,6,8a,8p,9,12a,12b,12c,12p,13,14a,14b,14c,16,17, according to the 2003 edition of lymph nodes group system defined by Japan Pancreas Society (JPS).
  Interventions: Procedure: resection of the nerve plexus on the right half of celiac and SMA associated with extended pancreatoduodenectomy
- pancreatoduodenectomy (Active Comparator): Standard pancreatoduodenectomy with regional lymph nodes includes group 5,6,8a,12b,12c,13,14a,14b,17, according to the 2003 edition of lymph nodes group system defined by Japan Pancreas Society (JPS).
  Interventions: Procedure: standard pancreatoduodenectomy

INTERVENTIONS:
Procedure: resection of the nerve plexus on the right half of celiac and SMA associated with extended pancreatoduodenectomy — Resection of the nerve plexus on the right half of celiac and SMA associated with extended pancreatoduodenectomy. Regional lymph nodes includes group 5,6,8a,8p,9,12a,12b,12c,12p,13,14a,14b,14c,16,17, according to the 2003 edition of lymph nodes group system defined by Japan Pancreas Society (JPS).
  Arms: pancreatoduodenectomy & nerve resection
Procedure: standard pancreatoduodenectomy — Standard pancreatoduodenectomy with regional lymph nodes includes group 5,6,8a,12b,12c,13,14a,14b,17, according to the 2003 edition of lymph nodes group system defined by Japan Pancreas Society (JPS).
  Arms: pancreatoduodenectomy

SUMMARY:
This study is performed to confirm whether resection of the nerve plexus on the right half of celiac and SMA associated with extended pancreatoduodenectomy could improve survival and relieve pain of pancreatic cancer patients.

DETAILED DESCRIPTION:
Lymph node metastasis and nerve invasion are characteristics of pancreatic cancer. For pancreatic head cancer, celiac and SMA nerve plexus are often involved. Many surgeons started to improve the surgical approach of pancreatoduodenectomy by extending the extent of surgical resection including an extended lymph node dissection and nerve plexus clearance in the hope of achieving better long-term survival rate. Postoperative complications such as diarrhea and malnutrition were reported after celiac and SMA nerve plexus resection during pancreatoduodenectomy. As a result, resection of the nerve plexus on the right half of celiac and SMA associated with extended pancreatoduodenectomy was recommended. This study is performed to confirm whether resection of the nerve plexus on the right half of celiac and SMA associated with extended pancreatoduodenectomy could improve survival and relieve pain of pancreatic cancer patients.

Subjects undergoing surgery will be randomized to extended pancreatoduodenectomy with resection of the nerve plexus on the right half of celiac and SMA versus standard pancreatoduodenectomy. Subjects will be followed every two months for survivorship or death to assess pain, quality of life measures, and narcotic pain control usage. The primary endpoint of overall survival and the secondary endpoint of disease-specific free survival will be determined at two year post surgery.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed content obtained prior to treatment
* Age ≥ 18 years and ≤ 80 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* The pathological staging does not exceed the stage IIB
* The expected survival after surgery ≥ 3 months
* Tumor locates at the head of the pancreas without distant metastasis
* No celiac trunk and superior mesenteric artery invasion by Loyer grading
* No operation contraindication

Exclusion Criteria:

* The pathological staging exceed the stage IIB
* Pancreatic cancer at the body and tail of the pancreas
* Benign tumor at the head of the pancreas
* Distant metastasis
* Severe important organ function impairment
* Active second primary malignancy or history of second primary malignancy within the last 3 years
* Pregnant or nursing women
* Human immunodeficiency virus (HIV)-positive patients
* Patients who are unwilling or unable to comply with study procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years

SECONDARY OUTCOMES:
Pain Control | 12 months
  Pain control will be assess by the Visual Analogue Scale (VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Pancreatic Cancer Institute, Shanghai, Shanghai Municipality, China